CLINICAL TRIAL: NCT05541393
Title: Engaging Church Health Ministries to Decrease COVID-19 (COVID-19) Vaccine Hesitancy in Underserved Populations in Baton Rouge
Brief Title: Engaging Church Health Ministries to Decrease Coronavirus Disease-19 Vaccine Hesitancy in Underserved Populations
Acronym: ENGAGE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant recruitment proved futile.
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 2021-047
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Education Group (Experimental): Participants randomized to the intervention will be engaged over a three-week period in discussions by their health ministries; any identified concerns or barriers around the initial vaccination series and/or booster vaccinations will be addressed and the importance of continued COVID-19 testing will be emphasized. Evidence-based vaccine strategies that focus on positive framing will be employed
  Interventions: Behavioral: Active Intervention Group
- Delayed Control Group (No Intervention): Participants in the delayed intervention control group will not receive any outreach during the three-week control period. Subsequent to completing the follow-up questionnaire, they will then be invited to join the intervention for the next three weeks. A follow-up questionnaire will be administered following their intervention period to be used in later analyses.

INTERVENTIONS:
Behavioral: Active Intervention Group — The intervention will involve meetings with the church health ministers to discuss COVID-19 vaccines and booster shots.
  Arms: COVID-19 Education Group

SUMMARY:
This study will determine the effectiveness of training church health ministers to educate their congregations about the safety and efficacy of COVID-19 vaccines and booster shots for decreasing vaccine hesitancy and improving testing knowledge in underserved Black communities.

DETAILED DESCRIPTION:
This study will determine the effectiveness of training church health ministers to educate their congregations about the safety and efficacy of COVID-19 vaccines and booster shots for decreasing vaccine hesitancy and improving testing knowledge in underserved Black communities. A total of 98 participants from three-to-five churches will be randomized to an intervention group that will receive counseling from their health ministers on the benefits of getting vaccinated, boosted, and tested, or to a delayed intervention control group. The effects of the intervention on the primary outcome, change in vaccine/booster hesitancy, will be assessed by a questionnaire that will be administered to both groups at baseline and after three weeks. Following the three-week control period, the delayed intervention control group will also receive the intervention and again be administered the questionnaire. Questionnaires will be used to obtain more granular information on sources of vaccine/booster hesitancy and for their vaccine-related decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y
* Not having received an initial COVID-19 vaccine or a booster vaccine at the recommended interval
* Having vaccine or booster hesitancy
* Able to understand and speak English
* Willing to engage with the church's health ministry via in-person or virtual/phone sessions

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in COVID-19 Vaccine/Booster Hesitancy from Baseline to 3 Weeks | Baseline and three weeks
  Vaccine hesitancy will be measured in those who indicate that they have not received the initial vaccine in a single or 2-series protocol using a single question: "How likely are you to get an approved COVID-19 vaccine?" Responses are recorded on a 7-point scale, with 1 being "not at all likely" and 7 being "very likely". Vaccine hesitancy will be defined as a score of 1 to 4 on the scale. Among individuals who have received the initial vaccine series, but not the booster, booster hesitancy will be measured using the following question: "How likely are you to get an approved COVID-19 booster shot?" Responses are recorded on a 7-point scale, with 1 being "not at all likely" and 7 being "very likely". Booster hesitancy will be defined as a score of 1 to 4 on the scale.

SECONDARY OUTCOMES:
Change in Vaccine/Booster Uptake from Baseline to 3 Weeks | Baseline and three weeks
  Change in vaccine or booster status

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified individual-level dataset will be made available to researchers making a reasonable request to the principal investigator. Data will be made available 1 year after publication of the primary outcomes manuscript.
Supporting Information: Study Protocol
Time Frame: Data will be made available 1 year after publication of the primary outcomes manuscript.
Access Criteria: Data will be available upon reasonable request.